CLINICAL TRIAL: NCT01844349
Title: Understanding the Nutritional Transition in the Maghreb to Contribute to the Prevention of Obesity and Non-communicable Diseases
Brief Title: Nutritional Transition in the Maghreb and Prevention of Obesity and Non-communicable Diseases
Acronym: Obe-Maghreb
Status: Completed | Type: Observational
Sponsor: Agnes GARTNER (Other Government)
Responsible Party: Sponsor-Investigator, Agnes GARTNER, Researcher, Institute of Research for Development, France
Organization: Institute of Research for Development, France (Other Government)
Other Study IDs: Corus 6028-2
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Iron Deficiency,; Anaemia,; Overweight,; Metabolic Syndrome
Keywords: North Africa; Urban women; Double burden of malnutrition; Iron depletion; Overweight/obesity; Metabolic syndrome; Abdominal obesity; Excess body fat
MeSH Terms: conditions — Iron Deficiencies; Anemia; Overweight; Metabolic Syndrome; Obesity; Obesity, Abdominal

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Problematic and state of the art Obesity and its associated non communicable diseases (NCDs) are rising rapidly in middle income countries, such as those in the Maghreb (North Africa). This progression is related to the context of a nutrition transition (changing food and physical activity environment) and profound changes in technological advances and in society. These societies and their health systems are insufficiently prepared for this evolution, which has enormous health and socioeconomic consequences. In the context of limited resources, the priority has been given on an international level to prevention. But several problems arise: - these countries are still confronted by undernutrition in terms of micronutrient deficiencies, which coexist with obesity and NCDs, including at a family level and also individual level. Known as the 'double burden', this coexistence is relatively new and has been rarely documented until recently. Educational measures could be ineffective in a society where cultural norms do not recognise obesity and where changes in lifestyle are possibly not seen as acceptable. As well as information about citizen's knowledge of risk factors, data on their perceptions and attitudes are indispensable. Policies that involve changing the 'obesogenic' environment that individuals occupy is a priority.

Objectives of the project Overall aim: to contribute to the development of preventive strategies for obesity and chronic NCDs in the context of a nutrition transition.

Specific objectives: characterise the nature and size of the double burden (obesity/undernutrition) in regions, families and individuals; estimate the prevalence of biological and behavioural risk factors; characterise the psycho-sociocultural determinants of behaviour.

ELIGIBILITY:
Inclusion Criteria:

* To live in the region of the capital city
* To give free informed consent

Exclusion Criteria:

* Pregnancy

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Residents of the region of the capital city
Sampling Method: Probability Sample
Enrollment: 8218 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Body mass index in kg/m² | baseline

SECONDARY OUTCOMES:
Serum ferritin in µg/L | baseline

OTHER OUTCOMES:
Blood pressure in mm Hg | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Gartner, PhD, Principal Investigator — Institute of Research for Development
Locations (2):
- Faculty of Sciences, Ibn Tofaïl University, Kenitra, Rabat-Salé, Morocco
- National Institute of Nutrition and Food Technology (INNTA), Tunis, Great Tunis, Tunisia

REFERENCES:
- [Derived] Ben Cherifa F, El Ati J, Doggui R, El Ati-Hellal M, Traissac P. Prevalence of High HDL Cholesterol and Its Associated Factors Among Tunisian Women of Childbearing Age: A Cross-Sectional Study. Int J Environ Res Public Health. 2021 May 20;18(10):5461. doi: 10.3390/ijerph18105461. PMID 34065252
- [Derived] Sassi S, Abassi MM, Traissac P, Ben Gharbia H, Gartner A, Delpeuch F, El Ati J. Intra-household double burden of malnutrition in a North African nutrition transition context: magnitude and associated factors of child anaemia with mother excess adiposity. Public Health Nutr. 2019 Jan;22(1):44-54. doi: 10.1017/S1368980018002495. Epub 2018 Oct 9. PMID 30298796
- [Derived] Traissac P, El Ati J, Gartner A, Ben Gharbia H, Delpeuch F. Gender inequalities in excess adiposity and anaemia combine in a large double burden of malnutrition gap detrimental to women in an urban area in North Africa. Public Health Nutr. 2016 Jun;19(8):1428-37. doi: 10.1017/S1368980016000689. Epub 2016 Apr 6. PMID 27049694
- [Derived] Gartner A, El Ati J, Traissac P, Bour A, Berger J, Landais E, El Hsaini H, Ben Rayana C, Delpeuch F. A double burden of overall or central adiposity and anemia or iron deficiency is prevalent but with little socioeconomic patterning among Moroccan and Tunisian urban women. J Nutr. 2014 Jan;144(1):87-97. doi: 10.3945/jn.113.178285. Epub 2013 Nov 6. PMID 24198310
- [Derived] Gartner A, Berger J, Bour A, El Ati J, Traissac P, Landais E, El Kabbaj S, Delpeuch F. Assessment of iron deficiency in the context of the obesity epidemic: importance of correcting serum ferritin concentrations for inflammation. Am J Clin Nutr. 2013 Sep;98(3):821-6. doi: 10.3945/ajcn.112.054551. Epub 2013 Jul 24. PMID 23885047